CLINICAL TRIAL: NCT06545292
Title: Microsampling to Facilitate Drug Monitoring of Oncolytics
Brief Title: Microsampling for Therapeutic Drug Monitoring of Oral Oncolytics in Oncology Patients
Acronym: MSTDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, dr. Tom van der Hulle, Medical Oncologist, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 86496
Record Dates: First submitted 2024-07-11; First posted 2024-08-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Drug Monitoring
MeSH Terms: interventions — Drug Monitoring

STUDY DESIGN:
Intervention Model Description: A single center prospective clinical validation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microsampling arm (Experimental): Patients who use an oral oncolytic will be asked to provide twelve microsamples obtained by finger prick:
  * 6 dried blood spots (DBS)
  * 6 volumetric absorptive microsampling (VAMS))
  Interventions: Diagnostic Test: Therapeutic drug monitoring with a dried blood spot and microatainer.

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring with a dried blood spot and microatainer. — Patients who use an oral oncolytic will be asked to provide four paired whole blood (WB) samples obtained by venapuncture.

SUMMARY:
The aim of the study is to perform a clinical validation of the analytical method for dried blood spot microsampling of cabozantinib, pazopanib, sunitinib, lenvatinib, imatinib, abiraterone, enzalutamide, nivolumab, ipilimumab, pembrolizumab, atezolizumab, bevacizumab or enfortumab vedotin. The secondary objective is to test the feasibility of home monitoring (microsampling TDM) of cabozantinib, pazopanib, sunitinib, lenvatinib, imatinib, abiraterone, enzalutamide, nivolumab, ipilimumab, pembrolizumab, atezolizumab, bevacizumab or enfortumab vedotin in oncology patients.

DETAILED DESCRIPTION:
Rationale: Oral targeted anti-cancer drugs are a relatively novel group of drugs with a complex pharmacological profile. Due to the high pharmacokinetic interpatient variability and advised fixed dose a wide variability in blood concentrations is seen in patients. Chances for individuals patients are high to be either underdoses (>30% of patients) or overdoses (>15%), which can lead to either decreased efficacy or severe side effects. In recent years, the development of monoclonal antibodies has changed the standard of care for treatment of many cancer types. While a small group of patients can have persisting efficacy, costs of monoclonal antibodies are extremely high. While no predictive biomarker has been established to predict response before treatment, recent research has shown clearance of immune checkpoint inhibitors varies over time and predicts early response. Therapeutic drug monitoring (TDM), based on measured drug levels, is a well-established method for personalized dosing of drugs. It has become part of standard of care when treating patients with oral antineoplastic agents. Currently, venous blood sampling is performed at the hospital. Home sampling of oral oncolytics by taking capillary blood samples by patients themselves provides many benefits. It could reduce the burden of extra blood sampling at the hospital and the need for additional phone calls afterwards for dose guiding. As of today, microsampling of immune checkpoint inhibitors is exploratory. Additionally, home sampling offers the possibility to collect multiple samples over a dose interval, and to base dose recommendation on AUC, rather than only on trough concentrations (Ctrough). To achieve this goal, clinical validation and implementations studies for microsampling are warranted.

Objective: The primary objective is to perform a clinical validation of the analytical method for dried blood spot microsampling of cabozantinib, pazopanib, sunitinib, lenvatinib, imatinib, abiraterone, enzalutamide, nivolumab, ipilimumab, pembrolizumab, atezolizumab, bevacizumab or enfortumab vedotin. The secondary objective is to test the feasibility of home monitoring (microsampling TDM) of cabozantinib, pazopanib, sunitinib, lenvatinib, imatinib, abiraterone, enzalutamide, nivolumab, ipilimumab, pembrolizumab, atezolizumab, bevacizumab or enfortumab vedotin in oncology patients.

Study design: A single center prospective clinical validation study. Study population: Patients treated in the LUMC with cabozantinib, pazopanib, sunitinib, lenvatinib, imatinib, abiraterone, enzalutamide, nivolumab, ipilimumab, pembrolizumab, atezolizumab, bevacizumab or enfortumab vedotin.

Intervention (if applicable): Patients who use an oral oncolytic will be asked to provide twelve microsamples obtained by finger prick (eight dried blood spots (DBS) and four wet blood samples in microtainer EDTA) and four paired whole blood (WB) samples obtained by venapuncture. The paired samples have to be obtained within 5 minutes of each other. Sampling will take place before the ingestion of the oral oncolytic (through concentration, Cthrough) and every hour for three hours after drug administration (C1, C2 and C3).

Patients who receive immune checkpoints inhibitors will be asked to provide eight microsamples obtained by finger prick (six DBS and two wet blood in microtainer EDTA) and two paired WB samples obtained by venapuncture. Sampling will take place just before infusion (Ctrough) and 15 minutes after the end of the infusion (Cinfusion+0.25) of the next cycle of immune checkpoint inhibitors. Microsampling collection will be performed using two different sampling devices, HemaXis DB 10 and Mitra Clamshell. Patients will be assisted by a research nurse with the sampling of the first spot, and the sampling of the remaining spots will be performed by the patient. In order to evaluate patient satisfaction with both DBS sampling devices, patients will receive two kits for home use of both HemaXis DB 10 and Mitra Clamshell. Patients will be asked to perform four blood trough concentrations at home, two with every device. After obtaining the fourth sample, patients will be asked to send the samples by post to the laboratory. In order to evaluate patient satisfaction with both DBS sampling devices, patients will be asked to fill the System Usability Scale (SUS).

Main study parameters/endpoints: The primary endpoint is the method agreement between whole blood sample (WBS) and DBS. The secondary endpoints are the success rate of DBS and the difference in SUS score between HemaXis DB 10 and Mitra Clamshell.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* 18 years of age or older;
* Using one or more of the following drugs: Cabozantinib, Pazopanib, Sunitinib, Lenvatinib, Imatinib, Abiraterone, Enzalutamide, Nivolumab, Ipilimumab, Pembrolizumab, Atezolizumab, Bevacizumab or Enfortumab vedotin

Exclusion Criteria:

* Not able to sample themselves using a finger prick

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Method agreement between whole blood sample (WBS) and bry blood spot (DBS). | All samples will be collected within 3 months
  Blood concentrations of the oral oncolytic will be obtained 0 to 3 hours after ingestion of the oral oncolytic. Blood concentrations of immune checkpoint inhibitors will be obtained 0 hours after infusion and 15 minutes after end of the infusion. Passing-Bablok analysis will be performed to investigate a linear relationship between WBS and DBS. Bland-Altman analysis will be performed to evaluate method agreement. Method agreement between WBS and DBS was defined as ≥67% of the samples between the range of 0.80 and 1.20 (with or without correction factor following Passing-Bablok analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided